CLINICAL TRIAL: NCT01393652
Title: A Phase I, Randomized, Placebo-Controlled, Dose Escalating Cross Over Study To Evaluate The Safety, Toleration, Pharmacokinetics And Pharmacodynamics Of PF-05105679 Under Fasted Conditions In Healthy Volunteers
Brief Title: Single Dose, Dose Escalation Healthy Volunteers Study Of PF-05105679
Acronym: SINGLE DOSE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: B3351001
Record Dates: First submitted 2011-05-23; First posted 2011-07-13 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-09

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics Safety Tolerability Pharmacodynamics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1: Experimental intervention: PF-05105679 or placebo (Experimental): Cohort 1
  Interventions: Drug: PF-05105679
- Cohort 2: Experimental intervention: PF-05105679 or placebo (Experimental): Cohort 2
  Interventions: Drug: PF-05105679
- Cohort 3: Experimental intervention PF-05105679 or placebo and (Active Comparator): Cohort 3
  Interventions: Drug: PF-05105679

INTERVENTIONS:
Drug: PF-05105679 — Subjects will receive single ascending doses of PF-05105679 or placebo to investigate safety/tolerability and pharmacokinetics of PF-05105679
  Arms: Cohort 1: Experimental intervention: PF-05105679 or placebo
Drug: PF-05105679 — Subjects will receive single ascending doses of PF-05105679 or placebo to investigate safety/tolerability and pharmacokinetics of PF-05105679
  Arms: Cohort 2: Experimental intervention: PF-05105679 or placebo
Drug: PF-05105679 — Subject will be randomized to a treatment sequence, and assigned to placebo, 2 separate single doses of PF-05105679 in the fasted state and to controlled-release Oxycodone 20 mg (positive control) , with at least one week wash-out between doses.
  Arms: Cohort 3: Experimental intervention PF-05105679 or placebo and

SUMMARY:
This is a two part study. The purpose of the first part (Part A) is the evaluation of the pharmacokinetics, safety and tolerability after single ascending dose of PF-05105679. The second part (Part B) of this study will focus on the exploratory pharmacodynamics of PF-05105679 using pharmacodynamics markers (cold detection) in healthy volunteers. The doses selected in Part B will have been administered previously in the Part A of the study.

ELIGIBILITY:
Inclusion Criteria:

Healthy Volunteers

Exclusion Criteria:

Standard Healthy Volunteers

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability. | 3 days
Pharmacokinetics of single doses of PF-05105679 as measured by plasma concentrations- Cmax, Tmax, half life, AUC last, AUC(0-24) and MRT | 3 days

SECONDARY OUTCOMES:
Average AUC2min VAS (cold pressor test) of PF-05105679. | 24 hours
Cold detection threshold (°C) of PF-05105679. | 24 hours
Cold pain threshold (°C) of PF-05105679. | 24 hours
Stimulus-response function to cold stimuli following menthol application. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- [Derived] Winchester WJ, Gore K, Glatt S, Petit W, Gardiner JC, Conlon K, Postlethwaite M, Saintot PP, Roberts S, Gosset JR, Matsuura T, Andrews MD, Glossop PA, Palmer MJ, Clear N, Collins S, Beaumont K, Reynolds DS. Inhibition of TRPM8 channels reduces pain in the cold pressor test in humans. J Pharmacol Exp Ther. 2014 Nov;351(2):259-69. doi: 10.1124/jpet.114.216010. Epub 2014 Aug 14. PMID 25125580
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3351001&StudyName=Single%20Dose%2C%20Dose%20Escalation%20Healthy%20Volunteers%20Study%20Of%20PF-05105679